CLINICAL TRIAL: NCT05931601
Title: Early Initiated Vasopressor Therapy vs. Standard Care of Primarily Fluid Therapy in Hypotensive Patients in the Emergency Department - A Pragmatic, Multi-center, Superiority, Randomized Controlled Trial
Brief Title: Early Initiated Vasopressor Therapy in the Emergency Department
Acronym: VASOSHOCK
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Lasse Paludan Bentsen, MD, Coordinating and Principal Investigator, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OP_1749; 2023-504584-16-00 (EU CTIS Number)
Record Dates: First submitted 2023-06-19; First posted 2023-07-05 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Shock; Shock, Septic; Hypotension; Hypotension and Shock; Hypotension Symptomatic; Hypovolemia; Hypovolemic Shock; Hypovolemic
Keywords: Peripherally infused noradrenaline; Fluid therapy; Fluid treatment; Non-hemorrhagic shock and hypotension; Emergency Department
MeSH Terms: conditions — Shock; Shock, Septic; Hypotension; Hypovolemia; Emergencies | interventions — Norepinephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Peripheral noradrenaline will be infused at rates of 0.05-0.15 mcg/kg/min for up to 24 hours after randomization in the ED until shock control is achieved.
  If shock control cannot be achieved, patients will be transferred to the ICU for further treatment of their condition but without further trial intervention.
  Weaning of intervention will be completed during the 24 hours, and if possible, terminated.
  If termination of treatment is not achievable within 24 hours, participants will be transferred to the ICU.
  Interventions: Drug: Noradrenaline
- Control (No Intervention): No ED administered noradrenaline. Standard care of hypotension and shock in the Danish ED's are fluid therapy and if not possible to achieve shock control, they are transferred to the ICU for administration of vasopressors if they are eligible for ICU admittance.

INTERVENTIONS:
Drug: Noradrenaline — See arm description
  Other Names: ATC-code C01CA03
  Arms: Intervention

SUMMARY:
The goal of this pragmatic, multi-center, superiority, randomized clinical trial is to compare early treatment with peripheral (through a vein) infused noradrenaline (a natural hormone that increases blood pressure) with fluid only therapy in patients with hypotensive and shock in the Danish and Swedish Emergency Departments (ED).

The main questions it aims to answer are:

If early initiated noradrenaline in non-bleeding hypotensive patients presenting in the ED can

* Improve time to shock control.
* Reduce the need for ICU admittance.
* Decrease mortality.

Participants will be included by the clinical staff and treated urgently with either noradrenaline or usual treatment during their Emergency Department stay.

After completion of the treatment in the Emergency Department, patient data will be extracted from the bed-side measurements, electronic health records and national registers.

Patients will be contacted by the research staff 1 year after study inclusion to answer brief questions about their daily physical function and ability to care for themselves.

Researchers will compare with patients receiving fluid therapy only, as this is the usual standard of care in Danish and Swedish Emergency Departments.

DETAILED DESCRIPTION:
Please refer to the full protocol.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Signs or suspicion of hypotension or shock (of any type such as septic, vasodilatory or hypovolemic not included in the exclusion criteria) defined as:

  1. SBP < 100mmHg or MAP < 65 mmHg combined with lactate > 2.0 mmol/L,
  2. Physician defined blood pressure for the individual patient combined with a lactate > 2.0 mmol/L
  3. Either SBP < 100mmHg or MAP < 65mmHg with obvious signs of shock with any lactate level evaluated by either two non-specialist physicians (e.g. registrar medical doctors) or a specialist physician.
* Received at least 500ml of intravenous fluid before study inclusion (Including prehospital administration) within the first 4 hours of ED arrival.
* Clinical Frailty Score (CFS) of ≤4. If CFS is ≥5 and the treating physician find the patient suitable for ICU admittance, the participant can be enrolled, if the on-call ICU doctor would accept the patient for ICU admittance. If the treating physician is unsure of ICU eligibility, regardless of CFS score, the patient should be consulted with the ICU consultant before study inclusion.

Exclusion Criteria:

* Cardiogenic, anaphylactic, haemorrhagic, or neurogenic shock suspected by the treating physician.
* Fertile women (<60 years of age) with positive urine human gonadotropin (hCG) or plasma-hCG or women breastfeeding.
* Patient deemed terminally ill or with a severe co-morbid status resulting in non-eligibility for ICU admittance decided by either the treating physician or ICU consultant.
* Known allergy to noradrenaline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2023-12-08 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is the proportion of patients achieving either SBP >100 mmHg or MAP > 65 mmHg or a target blood pressure set by the treating physician at 90 (±15) minutes after inclusion. | At 90 minutes
  Bed-side assessment during treatment and registered in the case report form.

SECONDARY OUTCOMES:
Number of intensive care unit (ICU) free days alive within 30 days | At 30 days
  Data is extracted from the Danish national registries or the patient's electronic medical record.
  Note: Death will count as 0 days.
Time without shock within 24 hours | At 24 hours
  Bed-side assessment during treatment and registered in the case report form or by extraction from the patient's electronic medical record.
30-day all-cause mortality | At 30 days
  Data is extracted from the Danish national registries or the patient's electronic medical records.
In-hospital all-cause mortality | At hospital discharge, an average of 30 days efter inclusion
  Data is extracted from the Danish national registries or the patient's electronic medical records.

OTHER OUTCOMES:
Proportion of patients receiving vasopressor at any point within 24 hours | At 24 hours
  Bed-side assessment during treatment and registered in the case report form or by extraction from the patient's electronic medical record.
Time to vasopressor initiation | At 30 days
  Bed-side assessment during treatment and registered in the case report form or by extraction from the patient's electronic medical record.
Hours of vasopressor infusion | At 30 days
  Bed-side assessment during treatment and registered in the case report form or by extraction from the patient's electronic medical record.
Proportion of patients with pulmonary oedema within 72 hours | At 72 hours
  Bed-side assessment during treatment and registered in the case report form or by extraction from the patient's electronic medical record.
Proportion of patients with acute kidney failure within 72 hours | At 72 hours
  Bed-side assessment during treatment and registered in the case report form or by extraction from the patient's electronic medical record.
Number of organ support free days alive within 30 days | At 30 days
  Organ support is defined as either mechanical ventilation, vasopressor/inotrope therapy or dialsysis.
  Data is extracted from the Danish national registries or the patient's electronic medical record.
Number of organ support free days alive within 30 days | At 30 days
  Organ support is defined as either mechanical ventilation, vasopressor/intotropic therapy or dialysis.
  Note: Death will count as 0 days.
  Data is extracted from the Danish national registries or the patient's electronic medical record.
Proportion of patients admitted to the ICU | At 30 days
  Data is extracted from the patient's electronic medical records.
ED Length of stay | At 72 hours
  Data is extracted from the patient's electronic medical records.
ICU length of stay | At 30 days
  Data is extracted from the patient's electronic medical records.
Hospital length of stay | At 30 days
  Data is extracted from the patient's electronic medical records.
Proportion and duration of mechanical ventilation | At 30 days
  Data is extracted from the patient's electronic medical records.
Proportion and length of renal replacement therapy | At 30 days
  Data is extracted from the patient's electronic medical records.
Amount of fluid therapy within the first 24 hours | At 24 hours
  Bed-side assessment during treatment and registered in the case report form or by extraction from the patient's electronic medical record.
Proportion of serious adverse events for noradrenaline or fluid therapy, e.g. extravasation or overdosis of noradrenaline, pulmonary edema, new cardiac arrhytmias, during the intervention of control period | At 24 hours
  Bed-side assessment during treatment and registered in the case report form or by extraction from the patient's electronic medical record.

CONTACTS AND LOCATIONS:
Overall Officials: Lasse P Bentsen, MD, Principal Investigator — Department of Emergency Medicine, Odense University Hospital; Mikkel Brabrand, MD, PhD, Study Chair — Department of Emergency Medicine, Odense University Hospital
Locations (8):
- Denmark (5):
  - Bispebjerg Hospital, Copenhagen
  - Esbjerg Hospital, Esbjerg
  - Gødstrup Regional Hospital, Herning
  - Zealand University Hospital, Køge
  - Odense University Hospital, Odense
- Sweden (3):
  - Department of Emergency Medicine, Helsingborg
  - Department of Emergency Medicine, Linköping
  - Department of Emergency Medicine, Ystad

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bentsen LP, Strom T, Forberg JL, Tiwald G, Biesenbach P, Kalmriz M, Rasmussen JH, Raaber N, Moller S, Lokke M, Tygesen GB, Nygaard H, Brok JH, Andersen JW, Bajusz N, Brabrand M. Early initiated noradrenaline versus fluid therapy for hypotension and shock in the emergency department (VASOSHOCK): a protocol for a pragmatic, multi-center, superiority, randomized controlled trial. Scand J Trauma Resusc Emerg Med. 2025 Apr 7;33(1):59. doi: 10.1186/s13049-025-01369-4. PMID 40197397
- See also: Related Info — https://www.kliniskforskning.dk/vasoshock/

DOCUMENTS (2):
  • Study Protocol (2024-12-09): https://cdn.clinicaltrials.gov/large-docs/01/NCT05931601/Prot_000.pdf
  • Statistical Analysis Plan (2025-06-15): https://cdn.clinicaltrials.gov/large-docs/01/NCT05931601/SAP_001.pdf